CLINICAL TRIAL: NCT01051713
Title: ENGAGED: E-Networks Guiding Adherence to Goals for Exercise and Diet
Acronym: ENGAGED
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Illinois Institute of Technology (Other)
Responsible Party: Principal Investigator, Bonnie Spring, Professor of Preventive Medicine, Psychology, and Psychiatry, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RC1DK087126-01 (NIH)
Record Dates: First submitted 2010-01-15; First posted 2010-01-18 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Obesity
Keywords: obesity; behavioraladherence; weight loss; smartphone
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard (Experimental): Those randomized to the Standard condition will record everything they eat and will total their daily fat grams and calories on the "Keeping Track" form used in the DPP. They will turn in their self-monitoring diaries and download their accelerometer (but not see those data) at weekly group sessions 1 through 8. Thereafter they will be expected to turn in paper data monthly, in person at the months 3 and 6 assessments and via mail, fax or e-mail for months 4 and 5. Accelerometer data will be downloaded at in-person visits.
  Interventions: Behavioral: Standard
- Technology Supported condition (Experimental): Those randomized to the Technology Supported condition will record dietary intake and weight on the smartphone, using the user-friendly, persuasive interface developed in Phase I. They will be expected to enter their dietary intake into the smartphone daily throughout the day. They will also be expected to enter their weight and to wear the accelerometer daily. Time-stamped data from the smartphone will upload automatically to the study server throughout the day, where it will be visible to the lifestyle coach. The participant's real-time diet, activity, and weight data relative to goals will also be visually depicted on the participant's smartphone. The anticipated web platform will be developed specifically for the ENGAGED participants. The coach will provide feedback on diet and activity self-monitoring and goal adherence at least weekly by phone, e-mail or text during weeks 1-8 and then at least monthly through the 6 month follow-up.
  Interventions: Behavioral: Technology Supported
- Self-Guided (No Intervention): Participants in the Self-Guided condition will receive DPP DVDs (3 DVDs and 1 CD) at the beginning of the study. This condition will not receive any direct dietary or physical activity interventions outside of the DVDs. Although Self-Guided participants will be receiving the same 7% weight loss goal as the other two groups, they will not be receiving physical activity or diet goals. The DVDs cover the initial 12-weekly sessions of the DPP, with the sessions portrayed by professional actors. They will also be provided with a supplemental DVD which includes a manual for each of the 12 sessions. They will also be giving the Keeping Track booklets and asked to record their diet and activity daily.

INTERVENTIONS:
Behavioral: Technology Supported — Those randomized to the Technology Supported condition will record dietary intake and weight on the smartphone, using the user-friendly, persuasive interface developed in Phase I. They will be expected to enter their dietary intake into the smartphone daily throughout the day. They will also be expected to enter their weight and to wear the accelerometer daily. Time-stamped data from the smartphone will upload automatically to the study server throughout the day, where it will be visible to the lifestyle coach. The participant's real-time diet, activity, and weight data relative to goals will also be visually depicted on the participant's smartphone. The anticipated web platform will be developed specifically for the ENGAGED participants. The coach will provide feedback on diet and activity self-monitoring and goal adherence at least weekly by phone, e-mail or text during weeks 1-8 and then at least monthly through the 6 month follow-up.
  Arms: Technology Supported condition
Behavioral: Standard — Those randomized to the Standard condition will record everything they eat and will total their daily fat grams and calories on the "Keeping Track" form used in the DPP. They will turn in their self-monitoring diaries and download their accelerometer (but not see those data) at weekly group sessions 1 through 8. Thereafter they will be expected to turn in paper data monthly, in person at the months 3 and 6 assessments and via mail, fax or e-mail for months 4 and 5. Accelerometer data will be downloaded at in-person visits.
  Arms: Standard

SUMMARY:
The ENGAGED study is a 12-month randomized controlled trial investigating different strategies to improve weight loss in overweight individuals. All participants will receive an effective weight loss treatment: either self-guided or group formats. All treatment will be provided in the Department of Preventive Medicine at Northwestern University. Participants who receive the self-guided weight loss treatment will be provided with a weight loss manual that contains proven behavioral weight loss strategies. Those participants who receive the group treatment will take part in 8 weekly, 90 minute group sessions in our clinic at 680 N. Lakeshore Dr., Chicago, IL 60048. Some participants will also be assigned an individual coach, who will communicate with them regularly via phone, email, and/or text message for the duration of the study. All participants must be willing and able to record food and beverage intake (either on a smartphone or on paper) and be willing to wear a small and unobtrusive physical activity measurement device for the first six-months of the study. Additionally, all participants will be asked to attend 3 follow-up assessment visits at our clinic at months 3, 6 and 12 after the study begins. Participants will be compensated for completing each of the 3 follow-up assessments. All participants will be part of a team weight loss competition at 3 and 6 months with financial incentive to be split evenly among the winning team.

DETAILED DESCRIPTION:
The Diabetes Prevention Program (DPP) intensive lifestyle intervention is the gold standard weight loss treatment for adults with cardiometabolic risk factors. Despite its efficacy, the DPP has not been widely adopted, because its 16 individual, face-to-face sessions with a specialist are considered too burdensome and expensive to be a sustainable program. Attempts to reduce cost by decreasing session number have yielded greatly diminished weight loss. Behavioral adherence to diet and activity goals declines and weight regain routinely begins once frequent face-to-face meetings cease. The still unmet challenge of DPP implementation is how to reduce treatment intensity without excising the regular social support, accountability, and feedback that are essential to maintain adherence. We hypothesize that it is feasible to implement DPP Intensive Lifestyle Treatment as effectively but twice as efficiently by using hand held technology to preserve feedback, accountability, and regular social support. The smartphone-based technology system to be tested is guided by Carver and Scheier's control systems theory of self-regulation. Initial formative research will upgrade the smartphone with engaging features that motivate participants to use the device to self-monitor and interact with a coach and peer support group. Use of the finalized tool will be compared to usual recording on paper records in a preliminary 3-group randomized controlled trial (RCT) involving 96 obese adults. By enabling peer support, accountability, and feedback on diet, physical activity, and weight loss goals continuously through the 6-month intervention period, the ENGAGED system is expected to enhance (1) behavioral adherence [operationalized by (a) self-monitoring of diet and activity and (b) attainment of diet and activity goals], and (2) weight loss. An enabling technology that integrates specialist and peer support resources to improve treatment adherence could help to curtail the obesity epidemic by increasing the efficiency, feasibility, and reach of effective DPP lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 30-40
* weight stable (not gained/lost more than 25 lbs in the past 6 months)
* not enrolled in any formal weight-loss program
* interested in losing weight
* willing and able to record dietary intake and weight for 6 months and wear an accelerometer
* willing to attend 8 weekly groups and 2 follow up assessments at the Northwestern Chicago campus
* expect to reside in the Chicago land area for the next 12 months

Exclusion Criteria:

* any unstable medical conditions (i.e. uncontrolled hypertension, diabetes, unstable angina pectoris, myocardial infarction, transient ischemic attack, cancer undergoing active treatment, a cerebrovascular accident within the past 6 months)
* history of insulin-dependent diabetes
* Crohn's disease
* diagnosis of obstructive sleep apnea requiring intervention
* required use of an assistive device for mobility (i.e. cane, wheelchair)
* BMI > 40
* hospitalization for a psychiatric disorder within the past 5 years
* those at risk for adverse cardiovascular events with moderate intensity activity
* those currently taking weight loss medication or committed to following an incompatible dietary regimen
* women who are pregnant, trying to get pregnant, or lactating
* Bulimia Nervosa
* suicide ideation
* current binge eating disorder
* those currently taking medications known to cause weight gain (i.e. Prednisone, Depakote, Diebeta, Diabinese, Cardura, Inderal, Zyprexa)
* current substance abuse or dependence
* plantar fasciitis
* current substance and/or alcohol dependence
* depression
* ADHD

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Weight loss | 3 months, 6 months, 12 months

SECONDARY OUTCOMES:
Behavioral adherence | 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, Ph.D., Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Spring B, Pellegrini CA, Pfammatter A, Duncan JM, Pictor A, McFadden HG, Siddique J, Hedeker D. Effects of an abbreviated obesity intervention supported by mobile technology: The ENGAGED randomized clinical trial. Obesity (Silver Spring). 2017 Jul;25(7):1191-1198. doi: 10.1002/oby.21842. Epub 2017 May 11. PMID 28494136
- [Derived] Pellegrini CA, Duncan JM, Moller AC, Buscemi J, Sularz A, DeMott A, Pictor A, Pagoto S, Siddique J, Spring B. A smartphone-supported weight loss program: design of the ENGAGED randomized controlled trial. BMC Public Health. 2012 Nov 30;12:1041. doi: 10.1186/1471-2458-12-1041. PMID 23194256